CLINICAL TRIAL: NCT03242499
Title: Lovastatin as a Neuroprotective Treatment for Early Stage Parkinson's Disease: a Single-center, Double-blind, Placebo-controlled Randomized Trial
Brief Title: Lovastatin as a Neuroprotective Treatment for Early Stage Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NCTRC201702
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Lovastatin 80mg per day for 48 weeks.
  Interventions: Drug: Lovastatin
- Placebo (Placebo Comparator): Placebo 80mg per day for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovastatin — Lovastatin 80mg or placebo use for 48 weeks.
  Other Names: LOVASTATIN "YUNG SHIN"
  Arms: Active
Drug: Placebo — placebo for 48 weeks
  Arms: Placebo

SUMMARY:
Background: Recent evidence has shown that statins, especially lipophilic statins, may have a neuroprotective benefit in Parkinson's disease (PD). We aim to perform a randomized placebo-controlled trial evaluating the disease-modifying efficacy of lovastatin in patients with early stage PD.

Methods and Study Design: This study will be a phase II, single-center, double-blind, randomized, placebo-controlled parallel-group study. In this trial, we are going to examine the possibility that lovastatin, a highly potent lipophilic statin, has disease-modifying effects in PD. We are going to enroll 80 patients with early stage PD patients. Subjects will then be randomized to a 48-week double-blind treatment period of lovastatin 80mg/day or placebo. Primary endpoints are changes in motor severity based on Movement Disorder Society-Unified Parkinson's Disease Rating Scale motor sub-score (MDS-UPDRS part III, with higher numbers indicating more severe disease). During the follow-up period, the dose of anti-parkinsonism could be added if both the patients and doctors thought the clinical condition deteriorated. Changes in PD medication as measured by levodopa-equivalent dose (LED) will be recorded at each visit. The secondary endpoints measured include MDS-UPDRS total scores, Part I and Part II sub-scores, the timing and dose of added anti-parkinsonism medication during the treatment period, the changes of 18F-DOPA PET uptake and MMSE scores, and global impression scale (GCI) of patients and investigators at the end of the study.

Expected results: We hypothesize that lovastatin would slow down both motor and cognitive symptoms deterioration and dopaminergic neuronal degeneration in patients with early stage PD.

Importance of the study: Our study will provide Class II evidence that intensive lipid lowering with lovastatin 80 mg/day decrease the disease progression in patients with early stage PD.

DETAILED DESCRIPTION:
This is a Phase 2, single-center, randomized, double-blind, placebo-controlled, parallel-group, 2-arm study in patients with mild to moderate PD. There will be three phases to the study. An initial 12-week screening phase was performed to determine eligibility. After informed consents, early-stage PD patients with Hoehn-Yahr stage 1 will be enrolled and participants will be asked to stop previously used anti-parkinsonism medications for at least one month to see the baseline disease severity. At the start of the study, participants will receive a comprehensive parkinsonism symptoms evaluation using Movement Disorder Society-Unified Parkinson's disease rating scale (MDS-UPDRS), global cognitive test using MMSE, and will be arranged for 18F-DOPA PET scan to evaluate the dopaminergic reserve in the striatum. Participants will also be asked to fasting for at least 8 hours to check the baseline laboratory test, including liver/renal functions, lipid profiles and serum CK level. Subjects will then be randomized to a 48-week double-blind treatment period of oral lovastatin 80mg/day or placeboSubjects in both groups will attend a further 5 clinic visits after 4, 12, 24, 36, and 48 weeks, where they are asked about their neurological symptoms and are evaluated by MDS-UPDRS. During the follow-up period, the dose of anti-parkinsonism could be added if both the patients and doctors thought the clinical condition deteriorated. Changes in PD medication as measured by levodopa-equivalent dose (LED) will be recorded at each visit. At final visit, patients will be arranged to receive the follow up 18F-DOPA PET scan to evaluate the dopaminergic reservation in the striatum and received MDS-UPDRS and MMSE evaluation. The secondary endpoints measured include MDS-UPDRS total scores, Part I and Part II sub-scores, the timing and dose of added anti-parkinsonism medication during the treatment period, the changes of 18F-DOPA PET uptake and MMSE scores, and global impression scale (GCI) of patients and investigators at the end of the study.

After informed consent form is completed, each patient will participate in the study for up to 48 weeks (a Screening Period of ≤12 weeks, followed by a Baseline Visit, 48 weeks of double-blind treatment, and a 4-week post-dose Safety Follow-up Visit) The post-dose Safety Follow-up Visit is for patients early terminating or not willing to participate in the open-label extension study):

* Screening Period: 16 weeks
* Treatment Period: 48 weeks
* Safety Follow-Up Period: 4 weeks After completion of the Treatment Period in this double-blind, placebo-controlled study, patients will be offered the option to enroll in an open-label extension study until 5 years. The end of the study is defined as the date of the last visit of the last patient in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is informed and given ample time and opportunity to think about his/her participation in this study and has given his/her written informed consent on an Independent Review Board (IRB) approved consent form.
* Patient is considered reliable and capable of adhering to the protocol, visit schedule, or medication administration according to the judgment of the investigator.
* Patient has a documented history of idiopathic PD consistent with the UK Parkinson's Disease Society Brain Bank Diagnostic criteria [14] prior to the Screening Visit.
* Modified Hoehn and Yahr stage =1 in the off medication state (stop medications for 1 month)
* Patients did not previously receive any anti-parkinsonism medications (drug naïve) or had stopped medications for at least 1 month.
* Age 30-90 years

Exclusion Criteria:

* Patient has any form of secondary or atypical parkinsonism (e.g., drug-induced, post stroke).
* Patient has known abnormality on brain CT or MRI imaging considered to be causing symptoms or signs of neurological dysfunction.
* Prior intracerebral surgical intervention for PD including deep brain stimulation (DBS).
* Prior or current use of statins as a lipid lowering therapy
* End stage renal disease (creatinine clearance eGFR <30 mL/min) or history of severe cardiac disease (angina, myocardial infarction or cardiac surgery in preceding two years)
* Abnormal liver function with aspartate transaminase (AST) or alanine transaminase (ALT) >2 x upper normal limit.
* Creatine kinase (CK) >2 x upper normal limit of normal.
* History of myopathy or rhabdolyolysis.
* Females who are pregnant or breast feeding.
* Patient has a history of chronic alcohol or drug abuse within the last 2 years.
* Exposure to neuroleptics (antipsychotic drugs) for more than 1 month within the past 2 years, or any exposure within the past year (except for quetiapine).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of MDS-UPDRS Part III (motor subscale) from baseline to week 48 | After informed consent form is completed, each patient will participate in the study for up to 48 weeks (a Screening Period of ≤12 weeks, followed by a Baseline Visit, 48 weeks of double-blind treatment, and a 4-week post-dose Safety Follow-up Visit
  Measure the motor symptoms severity changes of Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hsien Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No